CLINICAL TRIAL: NCT06503731
Title: A Global, Multicenter, Randomized, Double-Blinded, Placebo-Controlled, Phase 2 Study to Evaluate the Safety, Tolerability, and Efficacy of Efgartigimod PH20 SC Administered by a Prefilled Syringe in Kidney Transplant Recipients With Antibody-Mediated Rejection
Brief Title: A Study to Evaluate the Safety and Tolerability of Efgartigimod PH20 SC Given by Prefilled Syringe in Kidney Transplant Recipients With Antibody-Mediated Rejection (AMR)
Acronym: Shamrock
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2302; 2023-508180-72-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Antibody-mediated Rejection
Keywords: Active AMR; Chronic active AMR; Late AMR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment arm 1 (Experimental): Participants receiving Efgartigimod PH20 SC on top of optimized standard background immunosuppression therapy (tacrolimus, mycophenolate mofetil, and optionally steroids)
  Interventions: Combination Product: Efgartigimod PH20 SC - prefilled syringe
- Treatment arm 2 (Experimental): Participants receiving Efgartigimod PH20 SC on top of optimized standard background immunosuppression therapy (tacrolimus, mycophenolate mofetil, and optionally steroids) up to week 24 followed by placebo PH20 SC on top of optimized standard background immunosuppression therapy from weeks 24 to 48
  Interventions: Combination Product: Efgartigimod PH20 SC - prefilled syringe; Other: Placebo PH20 SC - prefilled syringe
- Treatment arm 3 (Placebo Comparator): Participants receiving Placebo PH20 SC on top of optimized standard background immunosuppression therapy (tacrolimus, mycophenolate mofetil, and optionally steroids)
  Interventions: Other: Placebo PH20 SC - prefilled syringe

INTERVENTIONS:
Combination Product: Efgartigimod PH20 SC - prefilled syringe — Subcutaneous efgartigimod PH20 SC given by prefilled syringe
  Arms: Treatment arm 1; Treatment arm 2
Other: Placebo PH20 SC - prefilled syringe — Subcutaneous placebo PH20 SC given by prefilled syringe
  Arms: Treatment arm 2; Treatment arm 3

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of efgartigimod PH20 SC given by a prefilled syringe in participants with Antibody-Mediated Rejection (AMR) after kidney transplantation.

After a screening period of up to 6 weeks, eligible participants will be randomized in a 1:1:1 ratio. The study drug will be administered subcutaneously while patients remain on their standard background immunosuppression therapy (tacrolimus, mycophenolate mofetil, steroids) during the treatment period (48 weeks). At the end of the treatment period, the participants will enter an observational/follow-up period (approximately 24 weeks). The participants will be in the study for up to 78 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant is within the ages of 18 and 80 years old
* The participant had a kidney transplant (living or deceased donor) at least 6 months before the study
* The participant has received a diagnosis of active or chronic active antibody-mediated rejection (AMR) with detectable donor-specific antibodies at time of the study
* A participant may be allowed into the study if they receive the following medications:

  1. Received mycophenolate mofetil for at least 20 weeks before the study
  2. Has remained on a stable dose of mycophenolate mofetil and tacrolimus for at least 4 weeks before being allowed to participate in the study
  3. Has remained on tacrolimus doses between 5 to 10 ng/mL at least 4 weeks before being allowed to participate in the study
  4. Steroid dose was between 0 to 10 mg per day of prednisone (or dose equivalent) for at least 4 weeks before being allowed to participate in the study

Exclusion Criteria:

* Confirmed T-cell or mixed rejection at time of the study
* Recent change in immunosuppressive therapy agents
* Any other medical condition that, in the investigator's opinion, would interfere with the results of the study or put the participant at undue risk
* Pregnant or lactating state or intention to become pregnant during the study

The complete list of criteria can be found in the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 78 weeks
Percentage of participants with permanent treatment discontinuation due to adverse events (AEs) | Up to 48 weeks

SECONDARY OUTCOMES:
Changes from baseline (slope) of the estimated glomerular filtration rate (eGFR) | Up to 72 weeks
Histological changes in kidney biopsy | Up to 72 weeks
Urine protein creatinine ratio (UPCR) | Up to 72 weeks
Graft and participant survival | Up to 72 weeks
Percentage change from baseline in total IgG levels in serum over time | Up to 60 weeks
Efgartigimod serum concentration-time profile and PK parameter Ctrough | Up to 48 weeks
Incidence of antidrug antibodies (ADA) against efgartigimod in serum over time | Up to 72 weeks
Incidence of antibodies against rHuPH20 in plasma over time | Up to 72 weeks

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Hospital, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Virginia Commonwealth University (VCU) Medical Center Hume-Lee Transplant Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Allgemeines Krankenhaus der Stadt Wien (AKH Wien) - Medizinischer Universitätscampus, Vienna, Austria
- Belgium (2):
  - Universitair Ziekenhuis (UZ) Gent, Ghent
  - Universitair Ziekenhuis Leuven (UZ Leuven) - Campus Gasthuisberg, Leuven
- London Health Sciences Centre, London, Canada
- Institut klinicke a experimentalni mediciny (IKEM), Prague, Czechia
- France (3):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire (CHU) de Grenoble Alpes - Hôpital Michallon, La Tronche
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hôpital de Rangueil, Toulouse
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Spain (4):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No